CLINICAL TRIAL: NCT01558115
Title: Denosumab in Primary Hyperparathyroidism
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAF2568; R01DK032333 (NIH); 20090741 (Other: Amgen)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Primary Hyperparathyroidism
Keywords: Columbia University; Primary hyperparathyroidism; Low bone density; Denosumab; Prolia
MeSH Terms: conditions — Hyperparathyroidism, Primary; Bone Diseases, Metabolic | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab - Group #1 (Experimental): Receive active drug for year 1 and year 2 of the study
  Interventions: Drug: Denosumab
- Placebo - Group #2 (Placebo Comparator): Receive placebo for year 1 and active drug for year 2 of the study
  Interventions: Drug: Denosumab; Other: Placebo

INTERVENTIONS:
Drug: Denosumab — The dose of denosumab is 60 mg every 6 months by subcutaneous injection.
  The 52 subjects will be randomly allocated (2:1) into treatment and placebo arms with the placebo group receiving a subcutaneous injection of vehicle in year 1. In year 2, those who were allocated to the study drug in year 1 will continue in year 2. Those who were allocated to placebo in year 1 will be crossed over to study drug in year 2.
  Group # 1: Receive active drug for year 1 and year 2 of the study
  Group #2: Receive placebo for year 1 and active drug for year 2 of the study
  Other Names: Prolia; Xgeva
Other: Placebo — The dose of denosumab is 60 mg every 6 months by subcutaneous injection. The placebo group will receive vehicle injections at the same time interval.
  The 52 subjects will be randomly allocated (2:1) into treatment and placebo arms with the placebo group receiving a subcutaneous injection of vehicle in year 1. In year 2, those who were allocated to the study drug in year 1 will continue in year 2. Those who were allocated to placebo in year 1 will be crossed over to study drug in year 2.
  Group # 1: Receive active drug for year 1 and year 2 of the study
  Group #2: Receive placebo for year 1 and active drug for year 2 of the study
  Arms: Placebo - Group #2

SUMMARY:
Primary hyperparathyroidism (PHPT), a disease characterized by excess parathyroid hormone (PTH) and high blood calcium, is one of the most common endocrine disorders. PHPT is seen most often in postmenopausal women. Many patients with PHPT have low bone mineral density (BMD) when bone mass is measured by dual energy x-ray absorptiometry (DXA), primarily at the forearm. There is currently no effective medical therapy which increases bone density at the forearm in patients with PHPT.

PTH both builds and breaks down bone, and the pathways by which PTH mediates these actions are beginning to be identified. Prior research suggests that RANKL, a molecule important in bone metabolism, responds to PTH, and that if the RANKL is inactivated, PTH is shifted towards building bone. The investigators will study the effect of Denosumab, a therapeutic agent that binds to and inactivates RANKL, in 28 postmenopausal women with PHPT. Our hypothesis is that Denosumab will increase bone mineral density in primary hyperparathyroidism.

The study will last two years, and subjects will be randomly assigned to receive either placebo or Denosumab for the first year of the study. In the second year, all subjects will receive Denosumab. Denosumab (60 mg) or placebo will be given every 6 months by an injection just under the skin. Study procedures performed will include bone mineral density tests by DXA, high-resolution peripheral quantitative computed tomography (HR-pQCT) scans, and assessments of biochemical markers of calcium metabolism and bone turnover using both blood and urine samples of subjects with PHPT.

DETAILED DESCRIPTION:
PTH has both catabolic and anabolic properties, and under normal circumstances, PTH in PHPT is catabolic for bone at the cortical skeleton. Recently, evidence for a direct role of PTH on RANKL expression and osteoclastogenesis in vivo was obtained using mice lacking a distant transcriptional enhancer of the RANKL gene that confers responsiveness to PTH. These observations, supported by additional cross-sectional studies in human subjects make a compelling argument that the catabolic actions of PTH are mediated by RANKL-mediated bone resorption.

The investigators now propose a proof of concept study to test the hypothesis that in PHPT, inhibition of the RANK-L pathway will unmask the anabolic potential of PTH. A therapeutic agent that redirects the actions of PTH in PHPT from one that is primarily catabolic to an anabolic one would fulfill this proof of concept. The investigators hypothesize that Denosumab, a human Immunoglobulin G (IgG) antibody that binds to and inactivates RANKL, will convert skeletal actions of PTH from catabolic to anabolic in primary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hypercalcemic PHPT in postmenopausal women with serum calcium >10.2 mg/dL and < 12.0 mg/dL (nl: 8.6-10.2)
* T-score between -1.5 and -2.5 at any site. If the T-score is <-2.5, patients become candidates for parathyroid surgery. They will be enrolled only if they refuse the parathyroid surgery

Exclusion Criteria:

* 25-hydroxyvitamin D level < 20 ng/ml
* Previous use of the bisphosphonate zoledronic acid (ever), alendronate or risedronate (within 12 months) or ibandronate (within 6 months)
* Current use of PTH, glucocorticoids, SERMS, estrogen (other than vaginal), calcitonin or pharmacological amounts of calcitriol Current or previous use of cinacalcet (within 6 months)
* Hyperthyroidism
* Rheumatoid arthritis or any other inflammatory joint disease
* Paget's disease of bone
* Malabsorption
* T-score <-3.5 at any site
* Signs of symptomatic PHPT (e.g, kidney stones within the past 5 years; fragility fracture within the past 2 years)
* Physical or mental handicapping condition that precludes ability to complete the protocol and/or provide informed consent.
* Subjects on Antiviral HIV therapy or subjects with compromised immune systems
* Premenopausal women or men
* Stage 5 Chronic Kidney Disease (CKD) or anyone on dialysis
* Creatinine clearance < 30 cc/min unless the patient is not a candidate for surgery or if the patient refuses surgery

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Bilezikian, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data were not collected per arm. This study was closed with the Institutional Review Board (IRB) in 2014 and additional analyses cannot be completed.
Groups:
- Denosumab - Group #1 or Placebo - Group #2: Denosumab - Group #1 Receive active drug for year 1 and year 2 of the study
  Placebo - Group #2 Receive placebo for year 1 and active drug for year 2 of the study
  Investigator is blinded
Period: Overall Study
Arm/Group | Denosumab - Group #1 or Placebo - Group #2
Started | 8
Completed | 1
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Study closed due to poor enrollment | 4

BASELINE CHARACTERISTICS:
Population: Study closed prematurely due to poor enrollment. The data were not collected per arm. This study was closed with the Institutional Review Board (IRB) in 2014 and additional analyses cannot be completed.
Arm/Group | Denosumab - Group #1 or Placebo - Group #2
Number analyzed (Participants) | 8
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 3
  > 65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) at the Lumbar Spine
Description: Percent change from baseline in BMD at the lumbar spine, as measured by Dual-emission X-ray absorptiometry (DXA) scan at 12 months
Time Frame: Baseline and 12 months
Population: Data was not collected and analyzed due to study closing prematurely because of poor enrollment.
Groups:
- Denosumab - Group #1: Receive active drug for year 1 and year 2 of the study
  Denosumab: The dose of denosumab is 60 mg every 6 months by subcutaneous injection.
  The 52 subjects will be randomly allocated (2:1) into treatment and placebo arms with the placebo group receiving a subcutaneous injection of vehicle in year 1. In year 2, those who were allocated to the study drug in year 1 will continue in year 2. Those who were allocated to placebo in year 1 will be crossed over to study drug in year 2.
  Group # 1: Receive active drug for year 1 and year 2 of the study
  Group #2: Receive placebo for year 1 and active drug for year 2 of the study
Arm/Group | Denosumab - Group #1 | Placebo - Group #2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Bone Mineral Density (BMD) at the Distal 1/3 Radius
Description: Percent change from baseline in BMD at the distal 1/3 radius, as measured by Dual-emission X-ray absorptiometry (DXA) scan at 12 months
Time Frame: 12 months
Population: Data was not collected and analyzed due to study closing prematurely because of poor enrollment.
Arm/Group | Denosumab - Group #1 | Placebo - Group #2
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Bone Mineral Density (BMD) at the Hip
Description: Percent change from baseline in BMD at the hip, as measured by Dual-emission X-ray absorptiometry (DXA) scan at 12 months
Time Frame: 12 months
Population: Data was not collected and analyzed due to study closing prematurely because of poor enrollment.
Arm/Group | Denosumab - Group #1 | Placebo - Group #2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: The data were not collected per arm. This study was closed with the Institutional Review Board (IRB) in 2014 and additional analyses cannot be completed.
Arm/Group | Denosumab - Group #1 | Placebo - Group #2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Data was not collected and analyzed as per protocol due to study closing prematurely because of poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes